CLINICAL TRIAL: NCT00197899
Title: Low-Dose Endotoxemia and the Acute Phase Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herlev Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KA 04015
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-12-13 (Estimated); Status verified 2005-09

CONDITIONS: Endotoxemia; Sepsis
MeSH Terms: conditions — Endotoxemia; Sepsis | interventions — endotoxin, Escherichia coli

INTERVENTIONS:
Drug: E. Coli endotoxin

SUMMARY:
The purpuse of this study is to examine the acute phase respons when different doses of E. Coli Endotoxin is injected in healty volunters.

ELIGIBILITY:
Inclusion Criteria: Healty volunteers -

Exclusion Criteria:

Infection 14 days prior to the trial Regular medication Present and /or former heart disease -

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2004-03; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, MD, DMSc, Study Chair — Department of Infectious Diseases 7641, University Hospital of Copenhagen, H:S Rigshospitalet; Dorthe H Olsen, MD, Principal Investigator — Department of Intensive Care, Herlev University Hospital; Dorthe H Olsen, DM, Study Director — Department of Intensive Care, Herlev University Hospital
Locations (1):
- Department of Intensive Care, Copenhagen, Copenhagen County, Denmark